CLINICAL TRIAL: NCT07384481
Title: Nursing Department Assistant Professor
Brief Title: Building Core Competencies of Taiwanese Care Food Specialists: Curriculum Design and Outcome Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: linchiahui
Record Dates: First submitted 2025-11-18; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Entrusted Professional Activities

STUDY DESIGN:
Intervention Model Description: hree-arm waitlist control trial (WCT) design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Student Immediate Intervention Group (IG): (Experimental): Students participated in the Core Competency Training Course for Eating Support Healthcare Aides, a 20-hour program designed to enhance knowledge and skills in providing safe and effective feeding support.
  Interventions: Other: Core Competency Training Course for Eating Support Healthcare Aides (20-Hour Course)
- Student Waitlist Control Group (WG) (Active Comparator): Student Waitlist Control Group (WG) Intervention:
  Participants in the Student Waitlist Control Group (WG) initially do not receive any training during the primary study period, serving as a delayed intervention control to account for time-related and external factors. After completion of all baseline and post-assessment measurements for the immediate intervention group (IG), the waitlist students then receive the same 20-hour Core Competency Training Course as the IG.
  Interventions: Other: Core Competency Training Course for Eating Support Healthcare Aides (20-Hour Course)
- Industry Group (RG) (Active Comparator): Industry Group (RG) Intervention:
  Participants in the Industry Group (RG) are current professional healthcare aides who receive the 20-hour Core Competency Training Course concurrently with the Student Immediate Intervention Group (IG). The timing ensures that the training is delivered during the same study period as the student intervention, allowing direct comparison of learning outcomes between students and experienced professionals.
  Interventions: Other: Core Competency Training Course for Eating Support Healthcare Aides (20-Hour Course)

INTERVENTIONS:
Other: Core Competency Training Course for Eating Support Healthcare Aides (20-Hour Course) — Core Competency Training Course for Eating Support Healthcare Aides, a 20-hour program designed to enhance knowledge and skills in providing safe and effective feeding support. The course comprised the following modules:
  1. Oral Changes and Basic Care Concepts (2 hours)
  2. Assisting Clients with Safe Eating (2 hours)
  3. Oral Hygiene and Care (3 hours, including practical skills)
  4. Dysphagia Diet Standards and Meal Texture Modification (2 hours)
  5. Food Storage, Cleaning, and Pre-/Mid-Processing (3 hours)
  6. Client Nutrition Knowledge (3 hours)
  7. Soft Food Selection and Preparation for Clients with Chewing Difficulties (2 hours)
  8. Hands-on Soft Food Preparation and Selection for Clients with Chewing Difficulties (3 hours)

SUMMARY:
Background: As Taiwan faces an aging population, the demand for long- term care services continues to rise, increasing the need for skilled care workers. Care Food Specialists, focusing on food preparation and oral health in long-term care, are essential for improving care quality.

Objective: This project aims to develop a core competency training curriculum for Care Food Specialists in Taiwan and assess its effectiveness in enhancing care worker skills.

Methods: Over two years, participants were recruited from various regions for training, with pre- and post-course assessments and qualitative interviews to evaluate changes in knowledge, attitude, and behavior.

Conclusion/Practical Applications: The project successfully designed and implemented a training curriculum, providing evidence of its positive impact on long-term care quality and offering a practical framework for future competency-based training.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of a Core Competency Training Course for Eating Support Healthcare Aides on knowledge and skills related to safe feeding practices, oral care, dysphagia diet management, and nutrition support for individuals with chewing or swallowing difficulties. The study employs a three-arm waitlist control trial (WCT) design, including both students and industry professionals, to comprehensively assess learning outcomes across different participant populations.

Study Design and Groups:

Participants are assigned to one of three groups:

1. Student Immediate Intervention Group (IG): Students receive the 20-hour training program at the beginning of the study.
2. Student Waitlist Control Group (WG): Students receive the same training after the initial study period, serving as a delayed intervention control.
3. Industry Group (RG): Current professional healthcare aides who receive the training concurrently with the student immediate intervention group.

This design allows comparison of pre- and post-intervention changes in the student immediate group, assessment of delayed intervention effects in the waitlist group, and evaluation of differences between students and industry professionals.

Participant Recruitment:

Student Group: Fifth-year junior college and third-year technical program students in long-term care-related programs, aged 19 years or older, who have completed a "Basic Care Practice and Laboratory" course and are able to attend the full 20-hour training. Students who are unwilling or have prior swallowing-related training are excluded.

Industry Group: Current professional healthcare aides aged 20 years or older with at least one year of experience in community or institutional long-term care settings, able to communicate in Mandarin and Taiwanese, and able to attend the full 20-hour course. Exclusion criteria include non-current employment, lack of language proficiency, or inability to complete the training.

Intervention (Training Program): The 20-hour Core Competency Training Course

Outcomes and Evaluation:

Participants' knowledge, practical skills, and competence in safe feeding and nutrition support are assessed pre- and post-intervention. Comparisons among groups allow evaluation of the training's immediate effects, delayed intervention impact, and differences between students and experienced professionals.

This comprehensive study design ensures both rigorous evaluation of the intervention's effectiveness and ethical inclusion of all student participants while providing practical insights for improving long-term care training programs.

ELIGIBILITY:
Student Group Inclusion Criteria

* Enrolled in a long-term care-related educational program (either a five-year junior college program or a four-year technical program).
* In the year immediately preceding graduation (fifth-year junior college students or third-year technical program students).
* Aged 19 years or older.
* Had completed the Basic Care Practice and Laboratory course.
* Able to attend the full 20-hour training course.

Exclusion Criteria:

* Unwilling to participate or unable to complete the full 20-hour course (e.g., due to other academic commitments)
* Industry Healthcare Aide Group

Inclusion Criteria:

* Currently employed as a professional healthcare aide in community-based or institutional long-term care settings.
* Actively working in a care aide role with at least one year of relevant experience.
* Possess a valid Taiwan Care Worker Training Certificate.
* Aged 20 years or older.
* Able to communicate in both Mandarin and Taiwanese.
* Able to attend the full 20-hour training course.

Exclusion Criteria:

* Younger than 20 years of age.
* Unable to communicate in Mandarin and Taiwanese.
* Not currently employed as a community or institutional care aide.
* Unable to complete the full 20-hour course

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Eating Support for Healthcare Aides (ESHA) Questionnaire | Baseline, Immediately after the 20-hour intervention course
  The scale is designed to assess caregivers' knowledge, attitudes, and behaviors regarding feeding and swallowing care. It was developed by Lin and Liu (2025) through literature review, expert Delphi consultation, and empirical testing, and comprises three domains with a total of 47 items.
  The knowledge domain includes 25 dichotomous items (correct/incorrect), with 1 point awarded for a correct answer and 0 points for an incorrect one; higher scores indicate more comprehensive knowledge. The reliability of this domain was examined using the KR-20 coefficient, yielding a value of 0.61. Item difficulty ranged from 0.60 to 0.99, and items demonstrated good discrimination, making the domain suitable as a baseline for comparing pre- and post-intervention educational outcomes.
  The attitudes and behaviors domains are assessed using a 5-point Likert scale, measuring caregivers' endorsement of feeding support and the frequency of its actual implementation, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Medical Foundation, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waldron C, Nunn J, Mac Giolla Phadraig C, Comiskey C, Guerin S, van Harten MT, Donnelly-Swift E, Clarke MJ. Oral hygiene interventions for people with intellectual disabilities. Cochrane Database Syst Rev. 2019 May 31;5(5):CD012628. doi: 10.1002/14651858.CD012628.pub2. PMID 31149734
- [Background] Newman R, Vilardell N, Clave P, Speyer R. Effect of Bolus Viscosity on the Safety and Efficacy of Swallowing and the Kinematics of the Swallow Response in Patients with Oropharyngeal Dysphagia: White Paper by the European Society for Swallowing Disorders (ESSD). Dysphagia. 2016 Apr;31(2):232-49. doi: 10.1007/s00455-016-9696-8. Epub 2016 Mar 25. PMID 27016216
- [Background] Chen S, Kent B, Cui Y. Interventions to prevent aspiration in older adults with dysphagia living in nursing homes: a scoping review. BMC Geriatr. 2021 Jul 17;21(1):429. doi: 10.1186/s12877-021-02366-9. PMID 34273953
- [Background] Lin CH, Liu MY. Development and Validation of the Eating Support for Healthcare Aides (ESHA) Questionnaire in Long-Term Care. Nutrients. 2025 Oct 15;17(20):3235. doi: 10.3390/nu17203235. PMID 41156487